CLINICAL TRIAL: NCT07154394
Title: Investigation of Cardiac Amyloid Deposits as a Cause of Cardiac Dysfunction in Alzheimer's Disease (Untersuchung Von Kardialen Amyloidablagerungen Als Ursache Einer Funktionseinschränkung Des Herzens Bei Alzheimer Demenz)
Brief Title: Cardiac Amyloid Deposits and Heart Dysfunction in Alzheimer's Disease
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Essen (Other)
Responsible Party: Sponsor
Other Study IDs: 20-9291-BO
Record Dates: First submitted 2025-05-20; First posted 2025-09-04 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2024-12

CONDITIONS: Dementia, Alzheimer Type; Mild Cognitive Impairment; Cardiac Amyloidosis
MeSH Terms: conditions — Alzheimer Disease; Cognitive Dysfunction; Amyloid Neuropathies, Familial

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients referred for cerebral amyloid PET to clarify Alzheimer's disease: The study population consists of patients who have been clinically referred for a cerebral amyloid PET examination to clarify a diagnosis of Alzheimer's disease.
  The study population will undergo a comprehensive diagnostic evaluation, which includes:
  * An extension of the amyloid PET examination to include cardiac PET/MRI imaging. No additional substances are applied and there is no additional radiation exposure.
  * A transthoracic echocardiogram, including strain analysis
  * A 12-lead electrocardiogram (EKG)

SUMMARY:
This study seeks to explore the possible common pathogenesis of both cardiac amyloidosis and Alzheimer's disease, which can both be associated with amyloid deposits. Using Positron Emission Tomography (PET) scans with amyloid tracers - a conventional tool for non-invasively imaging amyloid deposits in Alzheimer's disease - the research will extend this imaging methodology to the heart.

The study will conduct additional PET/MRI scans of the heart in patients undergoing amyloid tracer PET scans for Alzheimer's evaluations. Each participant will also undergo an echocardiogram and a clinical examination of dementia.

This could potentially enhance diagnostic practices in both cardiac amyloidosis and Alzheimer's disease.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing cerebral amyloid PET examination for clinical indication to clarify Alzheimer's disease
* No contraindications to undergo an MRI examination
* No contraindications to undergo an Amyloid PET scan

Exclusion Criteria:

* Patients with vascular dementia and confirmed other causes of dementia (e.g. stroke, vitamin deficiency, thyroid insufficiency, toxic causes such as alcohol)
* Patients with pronounced cardiac preconditions
* Pregnant and breastfeeding women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consists of patients who have been clinically referred for a cerebral amyloid PET examination to clarify a diagnosis of Alzheimer's disease.
  The study aims to recruit a diverse group of patients, aged 50-90 years, with a minimum of 7 years of education and good knowledge of the German language. Patients will be accompanied by a companion during the study.
  Excluded from the study will be patients with vascular dementia or other confirmed causes of dementia, such as stroke, vitamin deficiency, thyroid insufficiency, or toxic causes like alcohol. Additionally, patients with pronounced cardiac preconditions, pregnant women, and breastfeeding women will be excluded.
  The study population will be recruited from a clinical setting, where patients are undergoing routine diagnostic tests for Alzheimer's disease.
Sampling Method: Non-Probability Sample
Enrollment: 15 (Estimated)
Dates: Start 2022-08-15 (Actual); Primary Completion 2023-08-14 (Actual); Study Completion 2025-09-14 (Estimated)

PRIMARY OUTCOMES:
Frequency of occurrence of cardiac amyloid deposits in patients with a diagnosis of Alzheimer's disease (overall) | through study completion, an average of 1 year
Frequency of occurrence of cardiac amyloid deposits in relation to different disease manifestations (subdivided, for example, by clinical assessment of disease stage) | through study completion, an average of 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Essen, Essen, North Rhine-Westphalia, Germany

IPD SHARING:
Plan to Share IPD: No